CLINICAL TRIAL: NCT03783520
Title: Postoperative Pain After Using Er,Cr: YSGG Laser Irradiation Versus NaOCl Irrigation: A Randomized Controlled Clinical Trial
Brief Title: Postoperative Pain After Using Er,Cr,YSGG Lazer Irradiation During Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Görkem Özbilen, Specialist Dentist, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cukurova Endodontics
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Pain
Keywords: root canal treatment; intracanal irrigation; Laser
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Er,Cr:YSGG Laser (Experimental): In laser group, each root canal was dried with paper points and then Er,Cr:YSGG (Biolase™, Waterlase™, San Clemente, CA, USA) was used for intracanal disinfection with the following parameters: panel output power of 0,75 W, pulse frequency of 20 Hz, and 1% water pressure to 10% air pressure ratio laser with RFT3 tips (415 µm diameter radial firing tip RFT3 Endolase, Biolase Technology, Inc; calibration factor of 0.85). The fiber was placed at 1mm short of the WL. Irradiation was delivered along the entire length of the root canal with helicoradial movements, 1mm per seconds in speed. This procedure was repeated three times and kept for 20 seconds between each irradiation.
  Interventions: Device: Er,Cr:YSGG Laser
- Sodium hypochlorite (Active Comparator): In control group, each canal were irrigated with 6 ml of 2,5% NaOCl. For the final irrigation, 5 ml of sterile saline were used. During irrigation, needle was inserted 1 mm short of the WL.
  Interventions: Other: Sodium hypochlorite

INTERVENTIONS:
Device: Er,Cr:YSGG Laser — Er,Cr:YSGG Laser is used for disinfection of the root canals.
  Arms: Er,Cr:YSGG Laser
Other: Sodium hypochlorite — Sodium hypochlorite is used for disinfection of the root canals
  Arms: Sodium hypochlorite

SUMMARY:
Irrigation with sodium hypochlorite (NaOCl) during chemo-mechanic preparation for effective root canal disinfection is a standard protocol in root canal treatment. NaOCl is an alkali irrigant with pH 11.0 -12.0. Nearby its high antimicrobial efficacy, cytotoxic features make it questionable when it comes contact with periradicular tissues. Several irrigation materials were investigated less cytotoxic, more or equal antimicrobial to avoid such adverse effects. Calcium hypochlorite, chlorhexidine, chitosan and antibiotics are some of the chemicals tested. Laser is not a chemical but its action may show antibacterial effect. Studies showed that Er,Cr:YSGG laser is strongly antibacterial against Enterococcus faecalis biofilm. This antibacterial effect were frequently obtained with laser activated irrigation (LAI) or photon-induced photoacoustic streaming (PIPS) in the literature. The aim of this study was to evaluate whether disinfection procedure with laser provides more or less benefit in terms of postoperative pain when compared with the conventional NaOCl irrigation method.

DETAILED DESCRIPTION:
Both for maxillary and mandibular teeth, infiltration anesthesia were achieved by local anesthetic with 2 ml articaine hydrochloride with 1:200000 epinephrine (Maxicaine, VEM İlaç, Ist, Turkey). Endodontic access preparations were performed using diamond round burs. After the canals became visible, patency was checked with a K hand file (VDW, Munich, Germany), and a rubber dam was placed for isolation. The working length (WL) was determined with an electronic apex locator (Raypex 6, VDW) and accepted when three green bars were reached.

A crown-down preparation technique was performed using Reciproc nickel-titanium instruments (VDW, Munich, Germany) R#50 according to the manufacturers' instruction until the WL. During the instrumentation procedures, the root canals were irrigated with 6 ml of 2,5% NaOCl between each file.

In laser group, each root canal was dried with paper points and then Er,Cr:YSGG (Biolase™, Waterlase™, San Clemente, CA, USA) was used for intracanal disinfection with the following parameters: panel output power of 0,75 W, pulse frequency of 20 Hz, and 1% water pressure to 10% air pressure ratio laser with RFT3 tips (415 µm diameter radial firing tip RFT3 Endolase, Biolase Technology, Inc; calibration factor of 0.85). The fiber was placed at 1mm short of the WL. Irradiation was delivered along the entire length of the root canal with helicoradial movements, 1mm per seconds in speed. This procedure was repeated three times and kept for 20 seconds between each irradiation.

In control group, each canal were irrigated with 6 ml of 2,5% NaOCl. For the final irrigation, 5 ml of sterile saline were used. During irrigation, needle was inserted 1 mm short of the WL.

At the end of disinfection procedures, each root canal was dried with paper points and the largest gutta-percha cone that reached the WL without any resistance was used as the master cone. Measurements from the electronic apex locator were confirmed radiographically. In cases of discrepancies between the radiographic and electronic measurements, the latter was selected. All root canals were filled with gutta-percha and root canal sealer (Adseal Meta Biomed Co, Korea) using the lateral condensation technique. The teeth were coronally sealed with composite resin (Premise, Kerr, Salerno, Italy). After the completion of the root fillings, postoperative instructions were given to all patients and prescribed 200 mg ibuprofen only one tablet if it is needed within the 0- to 6-hour time interval after the treatment and then one for every 8 hours in the event of pain.

ELIGIBILITY:
Inclusion Criteria:

1)Single-rooted, maxillary and mandibular incisors, canines or premolars that were asymptomatic (no preoperative pain, swelling or acute endodontic or periodontal abscess). 2)Nonvital pulps and did not respond to cold testing.

3)People had no systemic diseases or allergies to local anesthetic agents . 4)People had not received any endodontic treatment previously. 5)People had no radiographic evidence of periapical bone loss.

Exclusion Criteria:

1. Pregnant and breastfeeding women
2. Patients taking analgesic, anti-inflammatory, or antibiotic medications during seven days prior to beginning of treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of Postoperative pain | 0-24 hours after root canal treatment
  Postoperative pain evaluation with verbal analog scale after root canal treatment. Patients signed as 0: no pain; 1: mild pain, analgesic not required; 2: moderate pain, analgesic required; 3: severe pain, analgesic has no effect in relieving the pain. The data were collected and statistically analysed using by the numerical data. In this study, "0" and "1" scores are considered as better outcome. Patients who signed these scores didn't need to use analgesics. The worst outcome is considered as the patients signed "3". Each scale range for each time interval evaluated as count of patient and presented as percentage. Scale ranges are not summed.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arias A, de la Macorra JC, Hidalgo JJ, Azabal M. Predictive models of pain following root canal treatment: a prospective clinical study. Int Endod J. 2013 Aug;46(8):784-93. doi: 10.1111/iej.12059. Epub 2013 Feb 12. PMID 23402273
- [Background] Dewsnup N, Pileggi R, Haddix J, Nair U, Walker C, Varella CH. Comparison of bacterial reduction in straight and curved canals using erbium, chromium:yttrium-scandium-gallium-garnet laser treatment versus a traditional irrigation technique with sodium hypochlorite. J Endod. 2010 Apr;36(4):725-8. doi: 10.1016/j.joen.2009.11.017. Epub 2010 Feb 6. PMID 20307752
- [Background] Figini L, Lodi G, Gorni F, Gagliani M. Single versus multiple visits for endodontic treatment of permanent teeth: a Cochrane systematic review. J Endod. 2008 Sep;34(9):1041-7. doi: 10.1016/j.joen.2008.06.009. PMID 18718362
- [Background] Christo JE, Zilm PS, Sullivan T, Cathro PR. Efficacy of low concentrations of sodium hypochlorite and low-powered Er,Cr:YSGG laser activated irrigation against an Enterococcus faecalis biofilm. Int Endod J. 2016 Mar;49(3):279-86. doi: 10.1111/iej.12447. Epub 2015 Apr 1. PMID 25772335